CLINICAL TRIAL: NCT02457390
Title: The Value of Contrast Enhanced Laparoscopic Ultrasound Examination During Robot-assisted Surgery for Primary Colorectal Cancer
Brief Title: The Value of CE-LUS During Robot-assisted Surgery for Primary Colorectal Cancer
Acronym: CE-LUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, MD Signe Bremholm Ellebaek, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140154
Record Dates: First submitted 2015-05-05; First posted 2015-05-29 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Cancer
Keywords: contrast enhanced laparoscopic ultrasound; CE-LUS; LUS; robot assisted CRC resection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CE-LUS (Experimental): Laparoscopic ultrasound examination (LUS) of the liver during robot assisted CRC surgery. The liver is systematically scanned for unrecognized liver metastases.
  After the laparoscopic LUS procedure, the liver is then systematically scanned with contrast enhancement with SonoVue® containing Sulphurhexafluoride. A bolus of 2.5 ml is injected into a peripheral vein followed by 10 ml of isotonic saline. The liver is then systematically scanned in 3 phases (arterial, venous and parenchymatous phase) searching for unrecognized liver metastases. The procedure is repeated after 5 minutes.
  The time it takes to do the scan is measured and any technical challenges are reported. Time, challenges and findings of liver metastases (number, segment and size) are entered on a registration form.
  Interventions: Procedure: CE-LUS

INTERVENTIONS:
Procedure: CE-LUS — To assess the use of contrast enhanced LUS during robot assisted primary CRC surgery. Does CE-LUS detect any unrecognized liver metastases.
  The patient will get a contrast-enhanced CT scan 3 month after surgery as a control to the CE-LUS procedure.
  Other Names: Sonovue

SUMMARY:
Laparoscopic ultrasound examination performed during surgery for primary cancer of the colon and rectum (CRC) has been shown to be able to detect liver metastasis that are not recognized by conventional computer tomography (CT scan) prior to surgery.

Today most of the colorectal cancer resections are performed by laparoscopy, but robotic technology is gradually developed in an attempt to overcome some of the limitations characterized by laparoscopy. The use of contrast enhanced laparoscopic ultrasound examination (CE-LUS) of the liver during robot-assisted CRC surgery has not been studied, and this despite the fact that it seems technically possible to perform.

With this project we will investigate whether CE-LUS associated with robotic surgery for CRC is technically feasible and whether it will be able to detect synchronous liver metastases that have not been detected on the preoperative imaging modalities.

DETAILED DESCRIPTION:
Title:

The value of contrast enhanced laparoscopic ultrasound examination during robot-assisted resection for primary colorectal cancer surgery.

Project:

The following project evaluates the value of contrast enhanced Laparoscopic Ultrasound examination (CE-LUS) in robot-assisted surgery for CRC.

The project "The value of contrast enhanced laparoscopic ultrasound examination during robot-assisted resection for primary colorectal cancer surgery" is a part of a Ph.D study at the University of Southern Denmark.

Purpose:

1.1: The primary purpose is to investigate whether the use of contrast enhanced ultrasound examination in connection with LUS procedure increases the number of detected liver metastases.

1.2: As a secondary objective; an evaluation of the technical feasibility of the CE-LUS procedure during robot-assisted resection for primary colorectal cancer surgery.

Background:

Laparoscopic surgery for cancer in the colon or rectum seems to be equal standing to open surgery with regards to the morbidity, mortality and the oncologic results (radicality and re-lapse frequency and long-term survival). Laparoscopic surgery for CRC is now a well-understood and well-established surgical method, but there are only few randomized trials dealing with the long-term results. The latest inventory work calls for better documentation of long-term results and calls for further randomized studies. Despite this, the number of laparoscopic operations for colorectal cancer (CRC) in Denmark is increasing, and laparoscopic surgery has become established as standard treatment for CRC. The development of minimally invasive surgery is not stopped by the laparoscopic approach, and robotic surgery is currently under evaluation in particular rectal surgery for CRC. Robot technology has been developed in an attempt to overcome some of the limitations that characterize the laparoscopic surgery. The establishment of a stable platform with instruments witch have increased rotating movements is an essential part of the robotic surgery. A motion-scaling and filtering makes sure that the image does not shake during the operation. The picture resolution is enhanced with 3D visualization and have visual magnification of the operating field. A combination of these features allows more precise dissection of tissue, suturing and improved bleeding-control compared to conventional laparoscopy.

Liver metastases are frequent in patients with CRC and about 15-20% of patients already have metastases at the diagnosis (synchronous metastases). Ultrasound examination during open surgery (IOUS) has shown to be an important diagnostic tool with high sensitivity (98%) and positive predictive value (86%) for detection liver metastases that are undiagnosed on preoperative CT or positron emission tomography (PET-CT). IOUS is considered as the gold standard for hepatic metastases within open surgery for CRC. In laparoscopic surgery this option disappears, but it is likely that laparoscopic ultrasound examination (LUS), may provide the same information as found by IOUS.

While laparoscopy and laparoscopic ultrasound examination (LUS) is well established in the staging and treatment of upper gastrointestinal cancers, this method is only sparsely evaluated in the treatment of CRC. There are only very few and older data dealing with the use of LUS in the TNM staging in patients with cancer in the colon and rectum. Several small studies have investigated the use of LUS to evaluate the M-stage in laparoscopic colorectal surgery and all studies show an increased detection of liver metastases. Overall, seems LUS to be better than the current pre-operative image modalities.

In prospective and blinded studies a percutaneous contrast-enhanced ultrasound examination (CEUS) of the liver proved to be able to detect significantly more liver-metastases from CRC than conventional percutaneous ultrasound.

With the new second-generation contrast agents CEUS seems to be equivalent to the contrast-enhanced CT and (magnetic resonance imaging) MRI for detection liver-metastases.

Liver metastases are frequent in patients with CRC and the use of intraoperative ultrasound (IOUS) during open surgery for CRC, has previously been regarded as the gold standard. Contrast-enhanced IOUS (CE-IOUS) during open surgery for CRC is only sparsely evaluated, but has been shown to increase sensitivity for detection liver-metastases.

Many patients with rectum cancer receive pre-treatment with chemotherapy and radiation therapy, and chemotherapy may make it difficult to identify existing metastases in the liver. Studies have shown an increased detection of metastases with contrast-enhanced ultrasound after pretreatment with chemotherapy.

The sensitivity of ultrasound examination can be improved by use of contrast enhanced ultrasound.There is a single pilot study dealing with contrast-enhanced laparoscopic ultrasound (CE-LUS) during primary CRC resection and the study revealed an improved detection of metastases.

In the same manner as in the laparoscopic resection of CRC, there is a need in the robot- assisted surgery to be able to compensate for the lack of intraoperative palpation and IOUS. The use of CE-LUS associated with robotic surgery in CRC patients has not been studied and this despite the fact that it appears technically possible to carry out the procedure for the robot procedure.

With this project we want to elucidate whether the use of CE-LUS in robot-assisted surgery for CRC will increases detection rate for liver metastases and evaluate the technical feasibility of the CE-LUS procedure.

Method:

The project is a prospective, descriptive study with 50 consecutive patients scheduled for robot-assisted surgery for primary CRC.

All patients had, prior to the scheduled surgery, completed a contrast enhanced CT of the chest and abdomen, as part of their Tumor, Lymph node and Metastases (TNM) evaluation. The CT scan was made according to current guidelines.

At the beginning of the surgery the patient will get the LUS examination by a specialist with skills in contrast-enhanced ultrasound. All liver segments are systematically scanned and any findings will be recorded on a registration form. After the LUS examination of the liver the procedure will supplied with a contrast enhanced examination. CE-LUS is performed with a contrast agent SonoVue® containing Sulphurhexafluoride which is a according to the department's instructions for CE-LUS procedure. A bolus of 2.5 ml is injected into a peripheral vein followed by 10 ml of isotonic saline. The liver is then systematically scanned in 3 phases (arterial, venous and parenchymatous phase) searching for unrecognized liver metastases. The procedure is repeated after 5 minutes.

The time it takes to do the LUS and CE-LUS is measured and any technical challenges are reported. Time, challenges and findings of liver metastases (number, segment and size) are entered on a registration form.

If there at the CE-LUS examination is found undiagnosed liver metastases, then the patient get an intraoperative LUS-guided fine-needle aspirations- biopsy (FNA) or tru-cut biopsy performed by a liver surgeon specialist and the lesion will be marked with a little silver pin. The latter is used for follow-up after pretreatment and to locate potential rest tumor. The patient will then be sent to the Department of Surgery A, Odense University Hospital, for a multidisciplinary tumor conference (MDT).

All other patients follow the Departments usual routines for adjuvant therapy. All patients included in the project will undergo a three-phase control CT scan 3 months after surgery. This is to evaluate whether there might be overlooked metastases during the CE-LUS evaluation.

All the information about the patients are entered and recorded in a database.

Ethics:

The project was reviewed and approved by the Science Ethics Committee, Project No:

S- 20140154. The project is reported to the Data Protection Agency. The studies will be registered in ClinicalTrials.com database. Participation in the project is voluntary, and patients may at any time withdraw their commitment to participation.

To date no reports of serious or life-threatening complications of LUS examinations or its probe is reported.

The LUS instrument/ probe is introduced into the abdominal cavity through the small holes ("gates") that the surgeon uses to do the operation with. Patients are not getting more scars / sores on the stomach than usual.

It is a specialist with expertise in ultrasound scanning, which handles the actual scan.

If there during the ultrasound scan is found spread of the cancer, which was not known before surgery, it may be necessary to take tissue samples from the suspicious area and perhaps mark this with a small silver pin. This is in order to regain these areas later, and to determine whether it is about the spread of cancer. In this case the patient will be further diagnosed and treated by the department's usual guidelines in this area.

The contrast agent used in this context is not associated with any serious risks and is a well-known and approved contrast agent. The ultrasound scan itself is not dangerous, and the contrast agent can give temporarily problems in form of headaches and nausea (prevalence 1-10%), and, rarely, transient weakness, vasodilation, hyperglycemia, sensory disturbances, rash and visual disturbances (frequency 0.1-1%). The contrast medium circulates only briefly in the body and the patient is monitored and are in general anesthetic, when administered. [26].

There is a minimal risk of bleeding in connection with a tissue sampling, but otherwise there are no side effects associated with the operation or construction of a small silver pin.

In the follow-up there is included an extra CT scan in relation to the department's usual procedure. There is a theoretical, but very modest risk- 0.01% in order to develop a new cancer disease.

Time and place The project is carried out at The RAK-Center at the department of Surgery A, Odense University Hospital, and the management at Department of Surgery A, Odense University Hospital, approves the project.

Schedule:

January 2015 - March 2016 : Inclusion of patients. March 2016 - September 2016: Data Processing and publications.

Project Manager:

MD PhD-student Signe Bremholm Ellebaek, Surgical Department A, Odense University Hospital

Other project participants:

Odense University Hospital, Surgical Department A. Professor, MD, PhD Michael Bau Mortensen MD PhD Claus W. Fristrup MD. Peiman Poornoroozy MD. Torsten Pless MD Bassam Mahdi, Radiology Department MD. Per V. Andersen

Economic Conditions:

There are sought financial support from various foundations, including the Cancer Society and the Region of Southern research funding, to conduct the study.

There are no commercial support givers, and the involved staff members get no financial gain.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to robot-assisted CRC resection
* patients with histologically verified cancer i colon or rectum
* informed consent
* patients with minimum age of 18
* patients without liver metastases

Exclusion Criteria:

* patients who have not given informed consent
* patients with severe heart disease, lung hypertension, or had had a heart attack < 7 days
* patients with alcohol or drug abuse.
* patients with liver metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Detection of synchronous liver metastases with CE-LUS | 3 months

SECONDARY OUTCOMES:
CE-LUS feasibility | 15 minuts
  CE-LUS feasibility will be assessed by a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Signe B Ellebaek, MD, Principal Investigator — Department of Surgery
Locations (1):
- Odense University Hospital, Odense, Odense, Denmark